CLINICAL TRIAL: NCT00805181
Title: Kinetics of Procalcitonin, C-reactive Protein and Pyuria in Uncomplicated Pyelonephritis in Women: A Pilot Study
Brief Title: Kinetics of Biomarkers in Acute Pyelonephritis
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Medical Director, University Hospital, Geneva
Other Study IDs: CER08-170; PRD-08-I-4
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Last update posted 2010-10-07 (Estimated); Status verified 2010-06

CONDITIONS: Pyelonephritis
MeSH Terms: conditions — Pyelonephritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute uncomplicated pyelonephritis

SUMMARY:
The objective of this study is to explore the kinetics of biomarkers in 30 adult female patients with uncomplicated acute pyelonephritis.

DETAILED DESCRIPTION:
We will measure c-reactive protein, procalcitonin, pyuria and a new blood biomarker (Signature TM) everyday till normalization of these markers in 30 adult female patients with uncomplicated acute pyelonephritis.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* Flank/loin pain or tenderness, or both and fever > 38°C during the last 48 hours and pyuria

Exclusion Criteria:

* Pregnancy
* Presence of indwelling catheters
* Known polycystic kidney disease or any malformation of the urinary tract, or single kidney; renal transplant recipients; acute or chronic renal failure requiring dialysis
* Recent discharge from hospital (during the last 10 days); ongoing antibiotic treatment
* Known severe immunosuppression: Receiver of solid-organ or hematopoietic stem cells transplants; neutropenia ( < 1 G neutrophils / L); chronic (more than 14 days) use of systemic glucocorticoids (>10 mg/d of prednisone); active use of immunosuppressive therapy for the treatment of auto-immune or inflammatory disease; HIV infection with < 350 CD4+ cells / ml or unknown CD4+ status
* Pyelonephritis initially identified as complicated: obstruction of urinary tract, urinary stone; history of renal infection in the last 15 days
* Patient with severe sepsis or septic shock

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 adult females with acute uncomplicated pyelonephritis
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2008-12; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Blood and urine biomarkers (procalcitonin, C-reactive protein, SIGNATURE(TM) test, pyuria | Daily till day 15.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier T Rutschmann, MD, MPH, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospitals, Geneva, Canton of Geneva, Switzerland